CLINICAL TRIAL: NCT00003019
Title: Vinblastine and Methotrexate in Children With Desmoid Tumor (Aggressive Fibromatosis) Which is Recurrent or Not Amenable to Surgical Resection or Irradiation - A Pediatric Oncology Group Phase II Study
Brief Title: Vinblastine and Methotrexate in Treating Children With Desmoid Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); Children's Cancer Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9650; POG-9650 (Other: Pediatric Oncology Group); CCG-P9650 (Other: Children's Cancer Group); CDR0000065601 (Other: Clinical Trials.gov); COG-P9650 (Other: Children's Oncology Group)
Record Dates: First submitted 2000-08-03; First posted 2004-04-30 (Estimated); Last update posted 2014-07-25 (Estimated); Status verified 2014-07

CONDITIONS: Desmoid Tumor
Keywords: desmoid tumor
MeSH Terms: conditions — Desmoid Tumors | interventions — Methotrexate; Vinblastine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Chemotherapy Treatment (Experimental): Patients receive vinblastine sulfate (5 mg/m2) IV and methotrexate (30 mg/m2) IV weekly for 26 weeks, then every 2 weeks for an additional 26 weeks. Treatment continues for a maximum of 1 year in the absence of unacceptable toxicity or disease progression. Patients with a complete response receive an additional 8 doses of chemotherapy. Patients are followed every 6 months for 4 years and then annually thereafter.
  Interventions: Drug: methotrexate; Drug: vinblastine sulfate

INTERVENTIONS:
Drug: methotrexate
  Other Names: MTX; amethopterin; NSC #000740
Drug: vinblastine sulfate
  Other Names: VBL; vincaleukoblastine; Velban; NSC #49842

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of chemotherapy with vinblastine and methotrexate in treating children who have desmoid tumors that are recurrent or untreatable with surgery or radiation therapy.

DETAILED DESCRIPTION:
OBJECTIVES: I. Estimate the efficacy and toxicity of vinblastine and methotrexate for newly diagnosed or recurrent desmoid tumors in children who are not good candidates for treatment with surgery or radiation therapy.

OUTLINE: Patients receive vinblastine and methotrexate IV weekly for 26 weeks, then every 2 weeks for an additional 26 weeks. Treatment continues for a maximum of 1 year in the absence of unacceptable toxicity or disease progression. Patients with a complete response receive an additional 8 doses of chemotherapy. Patients are followed every 6 months for 4 years and then annually thereafter.

PROJECTED ACCRUAL: A total of 13-25 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven, untreated, primary desmoid tumor (aggressive fibromatosis) for which surgery and/or radiation therapy is not thought to be feasible (prior attempted surgical resection allowed if gross residual disease remains) No other fibroblastic lesions or other fibromatoses allowed Recurrent desmoid tumor not previously treated with vinca alkaloids or methotrexate and no chemotherapy since recurrence Measurable disease by MRI

PATIENT CHARACTERISTICS: Age: Under 19 at time of diagnosis Performance status: Not specified Life expectancy: Not specified Hematopoietic: Hemoglobin normal for age WBC normal for age Platelet count normal for age Hepatic: Bilirubin less than 1.5 times upper limit of normal (ULN) for age SGOT less than 1.5 times ULN for age Renal: Creatinine less than 1.5 times ULN for age

PRIOR CONCURRENT THERAPY: See Disease Characteristics

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 28 (Actual)
Dates: Start 1997-08; Primary Completion 2003-07 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Event Free Survival
  To estimate the efficacy and toxicity of vinblastine and methotrexate for desmoid tumor in children with newly diagnosed or recurrent desmoid tumor who are not good candidates for treatment with surgery or radiation therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Steve Skapek, MD, Study Chair — St. Jude Children's Research Hospital; Bruce Himelstein, MD, Study Chair — Children's Hospital of Philadelphia
Locations (39):
- United States (36):
  - Long Beach Memorial Medical Center, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - David Grant Medical Center, Travis Air Force Base, California
  - Children's Hospital of Denver, Denver, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Children's Mercy Hospital, Kansas City, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - NYU School of Medicine's Kaplan Comprehensive Cancer Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Veterans Affairs Medical Center - Fargo, Fargo, North Dakota
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - Children's Hospital Medical Center - Cincinnati, Cincinnati, Ohio
  - Ireland Cancer Center, Cleveland, Ohio
  - Children's Hospital of Columbus, Columbus, Ohio
  - Doernbecher Children's Hospital, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Vanderbilt Cancer Center, Nashville, Tennessee
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
- Princess Margaret Hospital for Children, Perth, Western Australia, Australia
- Canada (2):
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - IWK Grace Health Centre, Halifax, Nova Scotia

REFERENCES:
- [Result] Skapek SX, Ferguson WS, Granowetter L, Devidas M, Perez-Atayde AR, Dehner LP, Hoffer FA, Speights R, Gebhardt MC, Dahl GV, Grier HE; Pediatric Oncology Group. Vinblastine and methotrexate for desmoid fibromatosis in children: results of a Pediatric Oncology Group Phase II Trial. J Clin Oncol. 2007 Feb 10;25(5):501-6. doi: 10.1200/JCO.2006.08.2966. PMID 17290057